CLINICAL TRIAL: NCT04407598
Title: Cross-Sectional Observation Telephone Survey Study to Understand the Changes in COPD Exacerbation Patterns and Potential Causes of These During the COVID-19 Pandemic
Brief Title: COPD in the Time of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0778
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-05

CONDITIONS: COPD Exacerbation; COPD
Keywords: COPD; AECOPD; COVID-19
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glenfield Complex COPD Clinic Cohort: Patients previously seen in the complex COPD clinic at the Glenfield Hospital.

SUMMARY:
This cross-sectional observational study will collect information about changes in exacerbation frequency and behaviour amongst a clinical cohort of severe or complex COPD clinic patients. This will be done through a combination of telephone survey and access to electronic heath records.

DETAILED DESCRIPTION:
This study will be a cross-sectional observational study utilising a telephone survey.

After obtaining informed verbal consent participants will be asked to recall their symptoms, exacerbation events and exacerbation medication usage over the periods of 01/03/20 - 14/03/20 (pre-lockdown) and then 15/03/20 to 30/04/20 (lockdown).

A structured survey will follow on from this asking questions regarding behaviour including self-isolation, shielding, other household contacts, visitors to the home, arrangements for shopping, changes in smoking behaviour (including that of other smokers in the household), medication changes, self-reported change in use of preventer medication, self-reported change in walking/activity levels and self-reported changes in anxiety levels.

Baseline clinical data will subsequently also be collected from the comprehensive respiratory review previously performed in the complex COPD clinic (comprising both hospital and GP records.) This will include previous AECOPD phenotyping (eosinophil levels, sputum culture and viral PCR), previous lung function testing, prescribed medication, BMI and smoking status and history. Previous AECOPD events will be counted and graded based on GP antibiotic or steroid prescriptions and hospital admissions.

Participants will be contacted once as part of the main study following verbal informed consent (via telephone). This will be a brief survey as described above, lasting approximately 20 minutes. A second similar survey will take place up to 12 months after the initial contact to evaluate longitudinal changes associated with the lockdown (further details on this will be submitted as an amendment at a later date due the shifting and unpredictable nature of the COVID-19 pandemic and lockdown, this will be prior to initiating these second calls).

Additional clinical data will be collected from healthcare records to quantify disease severity. Participant postcodes will be collected to link results with changes in local air pollution as recorded or estimated during the COVID-19 lockdown.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed clinical diagnosis of COPD
2. Ability to provide informed verbal consent via English language telephone consultation
3. Adults aged over 40 years

Exclusion Criteria:

1. Patients currently admitted to hospital
2. Unwilling/unable to provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients known to have COPD and previously seen in the Complex COPD Clinic at the Glenfield Hospital, Leicester.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in COPD Exacerbation Rate | 46 days
  The primary outcome will be the change in number of moderate or severe AECOPD events over the 46 days from the 15th March, 2020 to 30th April, 2020 compared to the same 46 day period in 2019.

SECONDARY OUTCOMES:
Change in number of Severe AECOPD events during period of interest in 2020 from same period in 2019. | 46 days
Change in Moderate AECOPD events during period of interest in 2020 from same period in 2019. | 46 days
Social contact changes during i) pre-lockdown and ii) lockdown period | 46 days
Household contacts during i) pre-lockdown and ii) lockdown period | 46 days
Household visitors during i) pre-lockdown and ii) lockdown period | 46 days
Regular shopping behaviour during i) pre-lockdown and ii) lockdown period | 46 days
Medication changes during i) pre-lockdown and ii) lockdown period | 46 days
Reported change in regular medication usage during i) pre-lockdown and ii) lockdown period | 46 days
Change in physical activity levels during i) pre-lockdown and ii) lockdown period | 46 days
Change in anxiety levels during i) pre-lockdown and ii) lockdown period | 46 days
Perceived fear of hospitalisation during COVID-19 period | 46 days
Patient reported changes in perception of symptoms, need for hospitalisation and availability and safety of healthcare resources thought semi-structured interviews in 20 patients (nested qualitative study) | 46 days
Association between changes in AECOPD event rate and changes in local air pollution during the COVID-19 lockdown | 46 days

CONTACTS AND LOCATIONS:
Overall Officials: Neil J Greening, PhD, Principal Investigator — University of Leicester
Locations (1):
- NIHR Leicester Biomedical Research Centre (Respiratory), Glenfield Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No